# CLINICAL STUDY DOCUMENT APPROVAL FORM

Study Name: Trevo Retriever Registry (China)

| Document Type: Statistical Analysis Plan (CDM10001420) | Document Date or Version: AA |
|---|---|
| We, the undersigned, have read and approve the d | We, the undersigned, have read and approve the document specified above: |
| 1. Name: Lixian Sun Functional Representative (FR) | Functional Role: BioStats Function Level: |
| Signature/Date: | 08/15/2018 |
| 2. Name: Yi-Ping Sun Functional Representative (FR) | Functional Role: CA Safety Function Level: |
| Signature/Date: 45 51 | 14 Aug 2018 |
| 3. Name: Dong Yu Manager (M) | Functional Role: CPM Function Level: |
| Signature/Date: | 8/14/2018 |
| 4. Name: | Functional Role: Choose an item. Function Level: select |
| Signature/Date: | · |
| 5. Name: | Functional Role: Choose an item. Function Level: select |
| Signature/Date: | |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

# Trevo® Retriever Registry (China)

Statistical Analysis Plan (SAP)

**Version AA** 

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

| Со | nter | | |
|----|----------|-------|--------------------------------------------|
| 1. | In | trod | uction3 |
| 2. | St | udy | Design |
| | 2.1. | St | tudy Objectives |
| | 2. | 1.1. | Primary Objective |
| | 2. | 1.2. | Secondary Objectives |
| | <br>2.2. | | tudy Endpoints |
| | | | • |
| | | 2.1. | Primary Endpoint3 |
| | 2. | 2.2. | Secondary Endpoints |
| 3. | Ar | nalys | is Population |
| 4. | Sa | ampl | e Size and Power |
| 5. | St | atist | ical Analysis |
| | 5.1. | P | rimary Endpoint |
| | 5.2. | | econdary Endpoints4 |
| | | 2.1. | Analysis Methods |
| | | | • |
| | | 2.2. | Secondary Endpoints Definition |
| | 5.3. | Α | dditional Safety Analyses5 |
| | 5.4. | D | escriptive Analyses5 |
| | 5. | 4.1. | Demographics and Baseline Characteristics5 |
| | 5. | 4.2. | Medical History5 |
| | 5. | 4.3. | Modified Rankin Scale (mRS)5 |
| | 5. | 4.4. | NIHSS |
| | 5. | 4.5. | Procedural Characteristics |
| | - | 4.6. | Device Malfunction |
| | | 4.7. | Time Intervals6 |
| | 5.5. | Sı | ubgroup Analyses6 |
| | 5.6. | Δ | d hoc Analyses |

Document Number: CDM10001420 Ver AA

6. Analyses Schedule

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

| 6. | Ana | lyses Schedule | . 6 |
|----|------|----------------------|-----|
| | 6.1. | Interim Analyses | . 6 |
| | 6.2. | Final Report | . 6 |
| 7. | Ana | lysis Software | . 6 |
| 8. | Ana | lysis Table Template | . 7 |

Document Title: Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### 1. Introduction

This document contains a detailed description of the Statistical Analysis Plan (SAP) for the data from the Trevo® Retriever Registry (China), coordinated with protocol of CDM 10001400.

This document provides specifications for the statistical analyses of the data to be analyzed for publications and presentations.

#### 2. Study Design

This Trevo® Retriever Registry is a prospective, open-label, multi-center, international trial. The purpose of the Trevo® Registry is to assess the performance of the Trevo® retriever in real world practice to increase knowledge on the performance of the device, monitor safety outcomes, detect rare complications, and to obtain information for potential improvements for next generation devices.

### 2.1. Study Objectives

### 2.1.1. Primary Objective

To assess real world performance of the CFDA cleared Trevo® Retriever intended to restore blood flow in the neurovasculature by removing thrombus in subjects experiencing ischemic stroke.

### 2.1.2. Secondary Objectives

- 1) To identify optimal interventional techniques, including type of anesthesia, access, and method of clot retrieval, to result in successful outcomes.
- 2) To provide robust registry data that maybe used to support expanded indications in regulatory submissions and support reimbursement dossiers.
- 3) To gather significant amount of real-world safety data to allow further subset analyses.

### 2.2. Study Endpoints

#### 2.2.1. Primary Endpoint

The primary endpoint is revascularization status at the end of the procedure using the modified TICI scale.

#### 2.2.2. Secondary Endpoints

- 1) Day 90 mRS (good clinical outcomes defined as mRS of 0-2).
- 2) Day 90 mortality.
- 3) Neurological deterioration at 24 hours.

Document Title: Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

4) Rates of device and procedure related Serious Adverse Events (SAE).

#### 3. Analysis Population

The Intent-to-treat principle will be followed to define the analysis population. All subjects who signed the informed consent and in whom Trevo® Retriever was deployed through the microcatheter are considered enrolled and will be included in all the analyses.

#### 4. Sample Size and Power

There will be no sample size/or power estimation for this single-arm registry. Two hundred subjects will be enrolled at up to 15 centers in China.

### 5. Statistical Analysis

#### 5.1. Primary Endpoint

Primary Endpoint is: Revascularization status at the end of the procedure.

The primary endpoint is measured using the modified TICI scale at the end of procedure. Success of primary endpoint was defined as a modified TICI score of 2b or better at the end of procedure.

Primary endpoint will be analyzed by percentages, frequencies and the 95% confidence interval of the percentage of success. The 95% confidence interval will be calculated using Clopper-Pearson exact method.

### 5.2. Secondary Endpoints

#### 5.2.1. Analysis Methods

Secondary endpoints will be analyzed by percentages, and frequencies.

#### 5.2.2. Secondary Endpoints Definition

- 1. Day 90 mRS (good clinical outcomes defined as mRS of 0-2).
- 2. Day 90 mortality.
  - If the subjects had completed their 90-day visit, the subjects will be considered as alive at Day 90. If the subjects did not come for their Day 90 visit and died, the date of death will be used to compare with the upper window of their Day 90 (90 + 14 days post procedure). If the subjects died after the upper window of their Day 90, the subjects will be considered as alive at their Day 90. Otherwise, the subjects will be counted as death before Day 90.
- 3. Neurological deterioration at 24 hours which is defined as four or more points increase in the NIHSS score from the baseline to 24 hours post procedure.

Document Title: Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

4. Rate of study device and procedure related serious adverse events (SAE) through Day 90.

### 5.3. Additional Safety Analyses

**Adverse Events** 

All SAEs through Day 90.

All SAEs through Day 90 will be summarized by number of events, number of subjects with events and the percentages of subjects with events by the type of SAEs and by their relatedness.

All AEs during procedure.

All AEs during procedure will be summarized by number of events, number of subjects with events and the percentages of the subjects with events by the type of AEs and by their relatedness.

### 5.4. Descriptive Analyses

### 5.4.1. Demographics and Baseline Characteristics

Subjects' demographic characteristics will be summarized using descriptive statistic methods.

Continuous variables will be summarized by mean±SD, median, minimum and maximum. Categorical variables will be summarized by percentages and frequencies.

#### 5.4.2. Medical History

Subjects' medical history will be summarized by percentages and frequencies.

#### 5.4.3. Modified Rankin Scale (mRS)

mRS will be summarized by frequencies and percentages and by visits. The difference of mRS from Day 90 to baseline, defined as mRS at Day 90 – mRS at baseline, will be categorized by decreased or no change (mRS from Day 90 - mRS from baseline<=0) or increased and will be analyzed by frequencies and percentages.

#### 5.4.4. NIHSS

NIHSS will be summarized by mean ± SD, median, minimum and maximum and by visits.

#### 5.4.5. Procedural Characteristics

The continuous variables will be summarized by mean ± SD, median, minimum and maximum. The categorical variables will be summarized by frequencies and percentages.

#### 5.4.6. Device Malfunction

All the device malfunction will be summarized by number of device malfunctions, number of device with device malfunction, percentage of device with device malfunction, number of subjects with device malfunctions and percentages of subjects with device malfunctions.

Document Title: Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### 5.4.7. Time Intervals

Time intervals will include but not limited to time from stroke symptom onset to admission to hospital/emergency department, intravenous tissue plasminogen (IV tPA), angio suite, arterial puncture, first Trevo® deployed, last Trevo® deployed and the end of the procedure. Time of clot integration, is calculated from the Trevo® deployed to the Trevo® starting to pulled.

### 5.5. Subgroup Analyses

Sub-group analyses (such as ICAD, IV Lytic use) for the Registry will be performed as needed.

### 5.6. Ad hoc Analyses

Ad hoc analyses will be generated as needed.

#### 6. Analyses Schedule

#### 6.1. Interim Analyses

Interim analysis may be performed as needed.

### 6.2. Final Report

Final report will be generated when all the 200 enrolled subjects complete their Day 90 visit or terminated before their Day 90.

### 7. Analysis Software

All statistical analyses will be generated using SAS® 9.4 or higher.

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

### 8. Analysis Table Template

The following tables are provided as samples and are subject to change as needed.

**Table 1 Subjects Disposition** 

| | Number of<br>Subjects<br>Enrolled<br>(N=xxx*) | Subjects Eligible at 24 Hours (- 6/+24) post procedure (N=xxx*) | Subjects Eligible at Discharge/Day 5-7 (whichever comes first) (N=xxx*) | Subjects<br>Eligible at<br>Day 30<br>(N=xxx*) | Subjects<br>Eligible at<br>Day 90<br>(N=xxx*) |
|---|---|---|---|---|---|
| Visit Completed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Visit Not Completed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reason for not completing the visit | | | | | |
| Missed Visit | NA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Early<br>Termination | NA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| List Reason for<br>Early Termination** | NA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>\*:</sup> N = Number of subjects expected at this visit

<sup>\*\*:</sup> The percentage is calculated based on the number of early terminations.

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

**Table 3: Baseline Demographics and Clinical Characteristics** 

| | Number of Subjects<br>(N=xxx) |
|---|---|
| Age | (IV-XXX) |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Gender | raun (raun, raun, |
| Male | xx.x% (xx/xxx) |
| Female | xx.x% (xx/xxx) |
| Body Mass Index | , , , |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Medical History | |
| Hypertension (HTN) | xx.x% (xx/xxx) |
| Heart Failure (CHF) | xx.x% (xx/xxx) |
| Coronary Artery Disease (CAD) | xx.x% (xx/xxx) |
| Extracranial Carotid Artery Disease | xx.x% (xx/xxx) |
| Left | xx.x% (xx/xxx) |
| Right | xx.x% (xx/xxx) |
| Bilateral | xx.x% (xx/xxx) |
| Atrial Fibrillation (A-fib) | xx.x% (xx/xxx) |
| Peripheral Vascular Disease (PVD) | xx.x% (xx/xxx) |
| Diabetes Mellitus | xx.x% (xx/xxx) |
| Other | xx.x% (xx/xxx) |
| Dyslipidemia | xx.x% (xx/xxx) |
| Current Smoker (within last year) | xx.x% (xx/xxx) |
| Past Smoker (>1 year ago) | xx.x% (xx/xxx) |
| Previous Transient Ischemic Attack (TIA) | xx.x% (xx/xxx) |
| Previous Ischemic Stroke | xx.x% (xx/xxx) |
| Previous Ischemic Stroke in the same erritory | xx.x% (xx/xxx) |
| Previous Intra-cerebral Hemorrhage | xx.x% (xx/xxx) |
| Previous History of known ICAD (intracranial | xx.x% (xx/xxx) |
| atherosclerotic disease) | |
| History of Alcohol Abuse | xx.x% (xx/xxx) |
| Other | xx.x% (xx/xxx) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### **Table 4: Baseline Lab**

| | Number of Subjects |
|------------------------|-----------------------|
| | (N=xxx) |
| Platelets (10^9/L) | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| PT (sec) | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| PTT (sec) | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| INR (RATIO) | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Blood Glucose (mmol/L) | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### **Table 5: Procedural Characteristics**

| | Number of Subjects<br>(N=xxx) |
|---|---|
| IA Medication Administered at Site of | xx.x% (xx/xxx) |
| Thrombus | *************************************** |
| Drug Type | |
| Lytic Used | xx.x% (xx/xxx*) |
| Anti-vasospasm | xx.x% (xx/xxx*) |
| Other | xx.x% (xx/xxx*) |
| Clot Location | rount (rogrout ) |
| CA - cervical | xx.x% (xx/xxx) |
| CA - petrous | xx.x% (xx/xxx) |
| ICA - cavernous | xx.x% (xx/xxx) |
| ICA - supraclinoid | xx.x% (xx/xxx) |
| ICAT bif | xx.x% (xx/xxx) |
| A1 | xx.x% (xx/xxx) |
| A2 | xx.x% (xx/xxx) |
| MCA-M1 | xx.x% (xx/xxx) |
| MCA-M2 | xx.x% (xx/xxx) |
| MCA-M3 | xx.x% (xx/xxx) |
| Vert | xx.x% (xx/xxx) |
| P1 | xx.x% (xx/xxx) |
| P2 | xx.x% (xx/xxx) |
| Target Vessel - Laterality | |
| Right | xx.x% (xx/xxx) |
| Left | xx.x% (xx/xxx) |
| Target Vessel Pass Basilar | |
| Proximal | xx.x% (xx/xxx) |
| Mid | xx.x% (xx/xxx) |
| Distal tip | xx.x% (xx/xxx) |
| Baseline Imaging | |
| CTP/CTA | xx.x% (xx/xxx) |
| MRI/MRA | xx.x% (xx/xxx) |
| Non-Contrast CT Only | xx.x% (xx/xxx) |
| Embolization to New Territory Observed | xx.x% (xx/xxx) |
| Distal Embolization Observed | xx.x% (xx/xxx) |
| Number Passes of Trevo® Retriever(s) | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

| Median (Q1-Q3) | xx.x (xx.x, xx.x) |
|---|---|
| Range (Min-Max) | xx.x (xx.x, xx.x) |
| 1 pass | xx.x% (xx/xxx) |
| 2 passes | xx.x% (xx/xxx) |
| >=3 passes | xx.x% (xx/xxx) |
| Number Passes of All Thrombectomy Device(s) | |
| Mean ± SD | xx.x ± xx.x (xxx) |
| Median (Q1-Q3) | xx.x (xx.x, xx.x) |
| Range (Min-Max) | xx.x (xx.x, xx.x) |
| *: Denominator is the number of subjects who used IA medicine | |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### **Table 6: Time Intervals**

| Time Intervals* | Number of Subjects<br>(N=xx) |
|-----------------------------------------------|------------------------------|
| Stroke symptom onset to first hospital | (ii Aliy |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to second hospital | , , , |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to primary hospital | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to IV Lytic | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to angiography suite | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to arterial puncture | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to first Trevo® deployed | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to last Trevo® deployed | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Stroke symptom onset to the end of procedure | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

| Range (min, max) | xx.x (xx.x, xx.x) |
|-------------------------------------|-----------------------|
| Stroke symptom onset to reperfusion | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Time of clot integration | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |

<sup>\*:</sup> Time intervals may be reported but not limited to those listed in the table. It will subject to change as needed.

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

Table 7: Modified Rankin Scale (mRS)

| Modified Rankin Scale (mRS) | % (n/N) |
|---------------------------------------------------|----------------|
| Pre-Stroke (N=xxx) | |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2 | xx.x% (xx/xxx) |
| Discharge/Day 5-7 (whichever comes first) (N=xxx) | |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2 | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 4 | xx.x% (xx/xxx) |
| 5 | xx.x% (xx/xxx) |
| 6 | xx.x% (xx/xxx) |
| 0-2 combined | xx.x% (xx/xxx) |
| Day 30 | |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2 | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 4 | xx.x% (xx/xxx) |
| 5 | xx.x% (xx/xxx) |
| 6 | xx.x% (xx/xxx) |
| 0-2 Combined | xx.x% (xx/xxx) |
| Day 90 | |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2 | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 4 | xx.x% (xx/xxx) |
| 5 | xx.x% (xx/xxx) |
| 6 | xx.x% (xx/xxx) |
| 0-2 Combined | xx.x% (xx/xxx) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

### **Table 8: Summary of NIH Stroke Scale (NIHSS)**

| NIH Stroke Scale (NIHSS) | Number of Subjects (N=xxx) |
|-------------------------------------------|----------------------------|
| Pre-procedure | |
| Mean ± SD (N) | xx.x ± xx.x (xxx) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| 24(-6/+24) post procedure | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |
| Discharge/Day 5-7 (whichever comes first) | |
| Mean ± SD (N) | $xx.x \pm xx.x (xxx)$ |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) |
| Range (min, max) | xx.x (xx.x, xx.x) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### **Table 9: Recanalization Results**

| Modified TICI | %(n/N) |
|---------------------------------------|--------------------|
| Subjects in Pre-procedure (N=xxx) | |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2a | xx.x% (xx/xxx) |
| 2b | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 2b+ | xx.x% (xx/xxx) |
| Subjects at the end of each pass* (N | I=xxx) |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2a | xx.x% (xx/xxx) |
| 2b | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 2b+ | xx.x% (xx/xxx) |
| Subjects at the end of procedure (N | I=xxx) |
| 0 | xx.x% (xx/xxx) |
| 1 | xx.x% (xx/xxx) |
| 2a | xx.x% (xx/xxx) |
| 2b | xx.x% (xx/xxx) |
| 3 | xx.x% (xx/xxx) |
| 2b+ | xx.x% (xx/xxx) |
| *: mTICI from all passes (up-to 6) ne | ed to be reported. |

### **Table 10: Primary endpoint**

| mTICI 2b+ at the end of procedure | % of subjects with mTICI2b+ | 95%CI |
|---|---|---|
| Yes | xx.x% (xx/xxx) | (xx.x%, xx.x%) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

### **Table 11: Secondary endpoints**

| Secondary Endpoints | % of Subjects with Clinical Outcomes (n/N)* |
|---|---|
| mRS** of 0-2 at Day 90 | xx.x% (xx/xxx) |
| Mortality rate at Day 90 | xx.x% (xx/xxx) |
| Neurological deterioration at 24(-6/+24) hours | xx.x% (xx/xxx) |
| Study Device and procedure related SAE | xx.x% (xx/xxx) |
| *:95% CI will be generated as needed for ad hoc analysis | |
| **: LOCF is used for Day 90 mRS. | |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

#### Table 12: All SAEs

| | # of events | Percentages of subjects with events* (Total subjects=xxx) |
|---|---|---|
| All SAEs | | |
| Details of all SAEs | xx | xx.x% (xx/xxx) |
| | xx | |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Study device and procedure related SAEs | | |
| Total | XX | xx.x% (xx/xxx) |
| Details of study device and procedure related SAEs | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| Study device related SAEs only | | |
| Total | XX | xx.x% (xx/xxx) |
| Details of study device related SAEs | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| Procedure but not study device related SAEs | | |
| Total | XX | xx.x% (xx/xxx) |
| Details of procedure but not study device related SAEs | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| Study device or procedure related SAEs | | |
| Total | XX | xx.x% (xx/xxx) |
| Details of study device or procedure related SAEs | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| Not study device and not procedure related SAEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details of not study device and not procedure related | xx | xx.x% (xx/xxx) |
| SAEs | | |
| | xx | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

Table 13: All AEs during procedure

| | # of events | Percentages of subjects with events* (N=xxx) |
|---|---|---|
| Total AEs | xx | xx.x% (xx/xxx) |
| Details of AEs during procedure | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Study device and procedure related AEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details of study device and procedure related SAE | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Study device related AEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details of study device related AEs | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Procedure but not study device related AEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details of procedure but not study device related AEs | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Study device or procedure related AEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details study device or procedure related AEs | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| Not study device and not procedure related AEs | | |
| Total | xx | xx.x% (xx/xxx) |
| Details of not study device and not procedure related SAEs | xx | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) |
| *: Some subjects may experience multiple events | | |

**Document Title:** Trevo® Retriever Registry (China) Statistical Analysis Plan

Document Number: CDM10001420 Ver AA

**Table 14: Device Malfunction** 

| | # of<br>events | Percentages of study<br>devices with events*<br>(Total device=xxx) | Percentages of subjects<br>with events**<br>(Total subjects=xxx) |
|---|---|---|---|
| Total | хх | xx.x% (xx/xxx) | xx.x% (xx/xxx) |
| Details of device malfunction | xx | xx.x% (xx/xxx) | xx.x% (xx/xxx) |
| | xx | xx.x% (xx/xxx) | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) | xx.x% (xx/xxx) |
| | XX | xx.x% (xx/xxx) | xx.x% (xx/xxx) |

<sup>\*:</sup> One device may have multiple malfunctions

<sup>\*\*:</sup> One subject may have multiple devices with malfunctions